CLINICAL TRIAL: NCT04766567
Title: Long Term Obstetric, Perinatal and Surgical Complications in Singleton Pregnancies Following Previous Cesarean Myomectomy
Brief Title: Complications in Singleton Pregnancies Following Previous Cesarean Myomectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bilge Hospital (Other)
Responsible Party: Principal Investigator, Oguz Guler, Principle investigator, Bilge Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1
Record Dates: First submitted 2021-02-01; First posted 2021-02-23 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Cesarean Section Complications
Keywords: Cesarean section; Cesarean myomectomy
MeSH Terms: interventions — Cesarean Section; Uterine Myomectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Serosal myomectomy (Experimental): Patients with singleton pregnancy, who had serosal myomectomy during cesarean section
  Interventions: Procedure: Cesarean section with cesarean myomectomy (serosal)
- Endometrial myomectomy (Experimental): Patients with singleton pregnancy, who had endometrial myomectomy during cesarean section
  Interventions: Procedure: Cesarean section with cesarean myomectomy (serosal)
- Control group (Placebo Comparator): Patients with singleton pregnancy, who did not have myomectomy during cesarean section
  Interventions: Procedure: Cesarean section without myomectomy

INTERVENTIONS:
Procedure: Cesarean section with cesarean myomectomy (serosal) — Serosal or endometrial myomectomy performed during cesarean section
  Other Names: Cesarean section with cesarean myomectomy (endometrial)
  Arms: Endometrial myomectomy; Serosal myomectomy
Procedure: Cesarean section without myomectomy — Cesarean delivery without performing myoemctomy
  Arms: Control group

SUMMARY:
The present study aims to investigate whether there is a difference in short- and long-term complications in patients undergoing cesarean myomectomy (endometrial or serosal myomectomy) during cesarean section.

DETAILED DESCRIPTION:
Myomectomy is frequently performed during cesarean section. Infertility, myoma recurrence, adhesions , uterine rupture (complete/incomplete), impaired uterine healing (partial or complete dehiscence/poor/good), placental abnormalities, and perinatal complications in subsequent pregnancy are may be associated with cesarean myomectomy. In this study, patients who underwent cesarean myomectomy during cesarean section in our institute were analyzed in a retrospective manner. Patients were divided into three groups as those receiving serosal myomectomy, endometrial myomectomy and those who only underwent cesarean section. The groups were compared with respect to the presence of adhesion formation, time to achieve pregnancy (fertility), morphology of the myomectomy scar, presence of uterine rupture and placental abnormalities.

ELIGIBILITY:
Inclusion Criteria:

* Participants should have singleton pregnancy delivered by cesarean section
* Cesarean section technique should include: Transverse hysterotomy to enter the uterine cavity, single layer closure of the uterine wall, non-sutured visceral and parietal peritoneum
* Myomectomy during cesarean section should include: only patients, who have undergone a single myomectomy and have been applied a single layer suture technique with the preservation of the pseudocapsule-for all cesarean myomectomy cases

Exclusion Criteria:

* Patients having history of any malignancy
* Patients with coagulation disorders
* Patients with a history of previous intraabdominal surgery on reproductive organs
* Patients with a history of endometriosis

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Complications of cesarean myomectomy | Post-cesarean 12 months
  The difference in the rate of complications associated with the cesarean myomectomy (presence of adhesion formation, time to achieve pregnancy (fertility), morphology of the myomectomy scar, presence of uterine rupture and placental abnormalities) in patients undergoing endometrial myomectomy, serosal myomectomy, or not receiving myomectomy during cesarean section

CONTACTS AND LOCATIONS:
Overall Officials: Oguz Guler, M.D., Principal Investigator — Bilge Hospital
Locations (1):
- Medicana Samsun Hospital, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No